CLINICAL TRIAL: NCT02861872
Title: Predictive Factors and Pharmacokinetics of Intra-peritoneal Chemotherapy
Brief Title: Intra-peritoneal Chemotherapy in Ovarian Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: MOGYN16IP
Record Dates: First submitted 2016-07-20; First posted 2016-08-10 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-07

CONDITIONS: Ovarian Neoplasms; Immune Tolerance; Neoplasms; Effects of Chemotherapy
Keywords: Ovarian; Ovarian cancer; Chemotherapy; Intraperitoneal chemotherapy; pharmacokinetics
MeSH Terms: conditions — Ovarian Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — EDTA blood and IP fluid
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- IP Patients: women, aged younger than 70 years, who will receive standard IP chemotherapy for advanced epithelial ovarian cancer, who are in an adequate physical and biochemical state to receive chemotherapy will be studied.

SUMMARY:
Ovarian cancer is the third most common gynecological malignancy worldwide. Because of late, aspecific symptoms, the disease is usually diagnosed at an advanced stage. Most patients experience recurrence and die as a result of the disease within 5 years. Treatment is a combination of surgical debulking and systemic administered chemotherapy. Intra-peritoneal (IP) chemotherapy with is currently considered the most effective treatment. In patients with at least an optimal surgical debulking, this leads to an improvement in life expectancy from 50 to 66 months. IP administration of chemotherapeutic agents is still not common practice. Furthermore recent studies revealed that cancer cells express a variety of tumor antigens, which can be targeted by the immune system. Also ovarian cancer shows evidence of a role for the immune system in clinical outcome. Novel insights into the mechanism of action of chemotherapy indicate that the efficacy of chemotherapeutic interventions are dependent on the modulation of the immune system. The impression exists that since IP chemotherapy is used, relatively more recurrences outside the abdominal cavity are observed. As of yet, no studies have described pharmacokinetics and pharmacodynamics of IP administered cisplatin and paclitaxel in the blood circulation. The investigators propose to study the use of this aspiration fluid from the IP cavity as a biomarker for the efficacy of chemotherapy intervention, monitor the effect of chemotherapy on IP tumor cells in the peritoneal cavity and monitor the effect of chemotherapy on immune cells present in the IP cavity. As well the investigators propose to correlate the presence and amount of tumor cells in peritoneal fluid with the debulking efficacy and CA 125 levels. Secondary to this the investigators intend to determine the pharmacokinetics of cisplatin and paclitaxel when administered in the IP cavity in the central circulation (plasma) as well as in the peritoneal fluid. In this observational explorative study women, aged younger than 70 years, who will receive standard IP chemotherapy for advanced epithelial ovarian cancer, who are in an adequate physical and biochemical state to receive chemotherapy are included. Immunological cell counts, tumor marker, immunological cell pathway activation and plasma concentrations of cisplatinum and paclitaxel in venous blood and in fluid aspirated from the abdominal cavity will be measured.

ELIGIBILITY:
Inclusion Criteria:

Patients receiving IP chemotherapy and therefore meeting the following criteria:

* Primary epithelial ovarian carcinoma FIGO stage III;
* Optimal or complete primary debulking (tumor rests ≤ 1cm;
* WHO 0 - 2;
* Adequate hematological function: WBC ≥ 3. 106/L en Platelets ≥ 100. 106/L,
* Adequate renal function (Creatinine clearance >60 ml/min (Cockcroft))
* Adequate liver function tests (bilirubin and/or transaminases <1.25 UNL)

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study (according to the standard IP chemotherapy):

* Intestinal stoma proximal to the flexura lienalis;
* Postoperative sepsis after primary debulking;
* Haemoglobin < 6.0 mMol/L
* Extended intraperitoneal adhesions;
* Neurotoxicity grade>1;
* Previous chemotherapy for ovarian carcinoma;
* Symptomatic hearing loss;
* Age >70 years.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women, aged younger than 70 years, who will receive standard IP chemotherapy for advanced epithelial ovarian cancer, who are in an adequate physical and biochemical state to receive chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Primary immunological endpoint: study the use of aspiration fluid from the IP cavity as a biomarker for the efficacy of chemotherapy intervention, measured by decrease in tumor cell count in IP fluid. | Change in tumor cell counts between samples 15 min before and after administration of chemotherapy through completion of chemotherapy during 18 weeks
Primary pharmacokinetic endpoint: study pharmacokinetics of cisplatin (platinum unbound fraction) when administered in the IP cavity in plasma and in the peritoneal fluid. | Change in platinum unbound fraction of cisplatin during the first course (first three weeks) of chemotherapy.
Primary pharmacokinetic endpoint: study pharmacokinetics of paclitaxel (plasma concentrations) when administered in the IP cavity in plasma and in the peritoneal fluid. | Change in plasma concentration of paclitaxel during the first course (first three weeks) of chemotherapy.

SECONDARY OUTCOMES:
Secondary immunological endpoint: rise in dendritic cells | Change in dendritic cell counts between samples 15 min before and after administration of chemotherapy through completion of chemotherapy during 18 weeks
Secondary immunological endpoint: rise in tumor infiltrating lymphocytes | Change in lymphocyte cell counts between samples 15 min before and after administration of chemotherapy through completion of chemotherapy during 18 weeks
Secondary immunological endpoint: rise in natural killer cells | Change in natural killer cell counts between samples 15 min before and after administration of chemotherapy through completion of chemotherpy during 18 weeks
Secondary immunological endpoint: decrease in macrophages M1 type | Change in macrophages M1 type cell counts between samples 15 min before and after administration of chemotherapy through completion of chemotherapy during 18 weeks
Secondary immunological endpoint: decrease in macrophages M2 type | Change in macrophages M2 type cell counts between samples 15 min before and after administration of chemotherapy through completion of chemotherapy during 18 weeks
Secondary immunological endpoint: change in cytokine level (IL-6) measured by ELISA | Change in IL-6 cytokine levels between samples 15 min before and after administration of chemotherapy through completion of chemotherapy during 18 weeks
Secondary immunological endpoint: change in cytokine level (IL-10) measured by ELISA | Change in IL-10 cytokine levels between samples 15 min before and after administration of chemotherapy through completion of chemotherapy during 18 weeks
Secondary immunological endpoint: change in cytokine level (IFNg) measured by ELISA | Change in IFNg cytokine levels between samples 15 min before and after administration of chemotherapy through completion of chemotherapy during 18 weeks
Secondary immunological endpoint: change in cytokine level (TNFa) measured by ELISA | Change in TNFa cytokine levels between samples 15 min before and after administration of chemotherapy through completion of chemotherapy during 18 weeks
Secondary immunological endpoint: change in cytokine level (CCL2) measured by ELISA | Change in CCL2 cytokine levels between samples 15 min before and after administration of chemotherapy through completion of chemotherapy during 18 weeks
Primary immunological endpoint: study the use of aspiration fluid from the IP cavity as a biomarker for the efficacy of chemotherapy intervention, measured by decrease in pSTAT in IP fluid. | Change in pSTAT between samples 15 min before and after administration of chemotherapy through completion of chemotherapy during 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nelleke Ottevanger, M.D. PhD., Study Chair — Internist-oncologist and principal investigator
Locations (1):
- Radboudumc, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Armstrong DK, Bundy B, Wenzel L, Huang HQ, Baergen R, Lele S, Copeland LJ, Walker JL, Burger RA; Gynecologic Oncology Group. Intraperitoneal cisplatin and paclitaxel in ovarian cancer. N Engl J Med. 2006 Jan 5;354(1):34-43. doi: 10.1056/NEJMoa052985. PMID 16394300
- [Background] Tewari D, Java JJ, Salani R, Armstrong DK, Markman M, Herzog T, Monk BJ, Chan JK. Long-term survival advantage and prognostic factors associated with intraperitoneal chemotherapy treatment in advanced ovarian cancer: a gynecologic oncology group study. J Clin Oncol. 2015 May 1;33(13):1460-6. doi: 10.1200/JCO.2014.55.9898. Epub 2015 Mar 23. PMID 25800756
- [Background] Schlappe BA, Mueller JJ, Zivanovic O, Gardner GJ, Long Roche K, Sonoda Y, Chi DS, O'Cearbhaill RE. Cited rationale for variance in the use of primary intraperitoneal chemotherapy following optimal cytoreduction for stage III ovarian carcinoma at a high intraperitoneal chemotherapy utilization center. Gynecol Oncol. 2016 Jul;142(1):13-18. doi: 10.1016/j.ygyno.2016.05.015. Epub 2016 May 21. PMID 27189456
- [Background] Wright JD, Hou JY, Burke WM, Tergas AI, Chen L, Hu JC, Ananth CV, Neugut AI, Hershman DL. Utilization and Toxicity of Alternative Delivery Methods of Adjuvant Chemotherapy for Ovarian Cancer. Obstet Gynecol. 2016 Jun;127(6):985-991. doi: 10.1097/AOG.0000000000001436. PMID 27159764
- [Derived] de Jong LAW, Lambert M, van Erp NP, de Vries L, Chatelut E, Ottevanger PB. Systemic exposure to cisplatin and paclitaxel after intraperitoneal chemotherapy in ovarian cancer. Cancer Chemother Pharmacol. 2023 Mar;91(3):247-256. doi: 10.1007/s00280-023-04512-z. Epub 2023 Mar 9. PMID 36892677